CLINICAL TRIAL: NCT00398385
Title: A Randomized Phase II Study of Preoperative Versus Postoperative Gemcitabine and Cisplatin for Patients With Stage IB-II Non-Small Cell Lung Cancer
Brief Title: Gemcitabine and Cisplatin Before or After Surgery in Treating Patients With Stage I or Stage II Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: NCC-NCCCTS-05-122; CDR0000516823 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2008-04

CONDITIONS: Lung Cancer
Keywords: squamous cell lung cancer; adenocarcinoma of the lung; adenosquamous cell lung cancer; bronchoalveolar cell lung cancer; large cell lung cancer; stage IB non-small cell lung cancer; stage IIA non-small cell lung cancer; stage IIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Gemcitabine; Chemotherapy, Adjuvant; Neoadjuvant Therapy

INTERVENTIONS:
Drug: cisplatin
Drug: gemcitabine hydrochloride
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving chemotherapy after surgery may kill any tumor cells that remain after surgery. It is not yet known whether giving chemotherapy before surgery is more effective than giving it after surgery in treating non-small cell lung cancer.

PURPOSE: This randomized phase II trial is studying gemcitabine and cisplatin to compare how well they work when given before or after surgery in treating patients with stage I or stage II non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the time to recurrence in patients with stage IB or II non-small cell lung cancer treated with neoadjuvant versus adjuvant gemcitabine hydrochloride and cisplatin.

Secondary

* Compare overall survival of patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.
* Compare quality of life of these patients.
* Compare the complete resection rate with and without neoadjuvant gemcitabine hydrochloride and cisplatin.

OUTLINE: This is a randomized study. Patients are stratified by disease stage (IB vs II) and histology (squamous cell carcinoma vs nonsquamous cell carcinoma). Patients are randomized to 1 of 2 treatment arms.

* Arm I (neoadjuvant chemotherapy): Patients receive gemcitabine hydrochloride IV over 30 minutes and cisplatin IV over 30 minutes on days 1 and 15. Treatment repeats every 4 weeks for up to 4 courses in the absence of disease recurrence or unacceptable toxicity. Within 8 weeks after initiating course 4 of chemotherapy, patients undergo complete surgical resection.
* Arm II (adjuvant chemotherapy): Patients undergo complete surgical resection. Beginning within 8 weeks after complete surgical resection, patients receive gemcitabine hydrochloride IV and cisplatin IV as in arm I.

Quality of life is assessed at baseline and periodically for up to 5 years.

After completion of study therapy, patients are followed periodically for at least 5 years or until disease recurrence.

PROJECTED ACCRUAL: A total of 170 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC)

  * Squamous cell or nonsquamous cell histology
* Stage IB or II disease
* Tumor amenable to curative surgical resection

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after completion of study therapy
* Medical fitness must be adequate for radical NSCLC surgery
* WBC ≥ 4,000/mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10 g/dL
* Bilirubin normal
* ALT and AST ≤ 2.5 times upper limit of normal
* Creatinine ≤ 1.5 mg/dL
* No second primary malignancy
* No active uncontrolled infection
* No concurrent serious disorder that would compromise patient safety or tolerance of study therapy
* No significant neurological or mental disorder
* No myocardial infarction within the past 6 months
* No symptomatic heart disease, including any of the following:

  * Unstable angina
  * Congestive heart failure
  * Uncontrolled arrhythmia

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or anticancer therapy
* No prior surgery for NSCLC
* No prior or concurrent radiotherapy or immunotherapy (e.g., biologic response modifier)
* No major surgery (other than biopsy) within the past 2 weeks
* No other concurrent anticancer therapy
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2005-05; Primary Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Time to recurrence

SECONDARY OUTCOMES:
Overall survival
Toxicity
Safety, in terms of frequency, severity, and relationship of adverse events, as assessed by NCI CTCAE v3.0
Complete resection rate
Quality of life as assessed by EORTC QLQ-C30 and EORTC QLQ-LC13 at baseline and periodically for 5 years
Patient population most at risk for disease recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Heungtae T. Kim, MD, PhD, Study Chair — National Cancer Center, Korea
Locations (1):
- National Cancer Center - Korea, Goyang, South Korea